CLINICAL TRIAL: NCT04778631
Title: Impact of Thermotherapy During Childbirth on Postpartum Perineal Pain: a Multicenter Factorial Randomized Controlled Trial
Brief Title: Impact of Thermotherapy During Childbirth on Postpartum Perineal Pain (PERISAFE)
Acronym: PERISAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Apicil (Other); PRIDE prize, Laboratoire Guigoz, Département Hopsitalo-universitaire Risques et Grossesse, Université de Paris (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP210326; 2020-A03399-30 (Other: ID-RCB Number)
Record Dates: First submitted 2021-01-24; First posted 2021-03-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pelvic Pain
Keywords: perineum; pelvic pain; acute pain; pain management; delivery; obstetric; labor stage; second; analgesia; obstetrical; postnatal care; heat therapy; cryotherapy
MeSH Terms: conditions — Pelvic Pain; Acute Pain; Agnosia; Neoplasm Metastasis; Hyperthermia | interventions — Diathermy; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Heat therapy (Experimental): Local perineal heat therapy during active second stage of labor
  Interventions: Device: Heat therapy
- Cryotherapy (Experimental): Local perineal cryotherapy during the immediate postpartum period
  Interventions: Device: Cryotherapy
- Active second stage usual car (No Intervention): Standard obstetrical care and perineal protection during active second stage of labor
- Postpartum usual care (No Intervention): Standard immediate (<2 hours) postpartum care

INTERVENTIONS:
Device: Heat therapy — Application of warm compresses, soaked in hot tap water (between 38° and 44 °C), to the perineum, at each contraction or pushing effort from the start of perineum distension until birth.
  Other Names: Warm compresses
  Arms: Heat therapy
Device: Cryotherapy — Application of a perineal instant col pack to the perineum, after placental delivery or perineum suturing, for at least 20 minutes.
  Other Names: Perineal instant coldpack
  Arms: Cryotherapy

SUMMARY:
Perineal pain is common after vaginal birth. Thermotherapy might be effective to limit postpartum perineal pain, thanks to the effects of local heating or cooling application. This study aims to evaluate the impact of thermotherapy during childbirth on postpartum perineal pain.

DETAILED DESCRIPTION:
Perineal lesions are common during vaginal delivery: 52% of women giving birth in France experience perineal lesions and 20% an episiotomy. Obstetrical anal sphincter injuries (OASIS) are the most feared due to the risk of anal incontinence, but they concerned a minority of women (0.8%). For most of the women with simple lesions of the perineum, the primary consequence is pain. This moderate to severe perineal pain affects between 40% and 95% of women and peaks in intensity the day after childbirth. This pain might be disabling, impair the mobility, the establishment of breastfeeding, the mother-infant bond, alter the emotional state and overall might affect the quality of life of mothers.

Thermotherapy provides a minimally invasive and inexpensive alternative to limit perineal pain in postpartum, thanks to the effects of local heating or cooling application to the perineum :

* Heat therapy with warm compresses, to protect the perineum during active second stage of labor and reduce the degree of perineal injury : the application promotes vasodilation and extensibility of tissues;
* Cryotherapy with instant cold pack, to prevent the onset of pain in the immediate postpartum period: the application limits the development of oedema or hematoma.

Midwives frequently use thermotherapy with heat or cold. However, these practices cannot be recommended due to a lack of data. Moreover, the potentially synergic effect of consecutive application of heat and cold therapy into the perineum during active second stage of labor and immediate postpartum period has never been evaluated. We hypothesize that thermotherapy during childbirth may reduce postpartum perineal pain.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women or multiparous women without history of vaginal birth
* singleton fetus
* fetal cephalic presentation
* ≥37 gestational weeks
* active labor (cervical dilatation ≥ 6 cm)
* living fetus
* major female Exclusion Criteria
* Abnormal fetal heart rate requiring hastening childbirth
* Fetal malformation, stillbirth
* History of female genital mutilation
* Women not understanding French
* Women with psychiatric condition
* Anonymous childbirth
* Minor female
* No affiliation to a social security scheme (beneficiary or assignee)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
Change of perineal pain assessed by the VAS (<H24) | From 2 to 24 hours after delivery
  Perineal pain intensity, as a mean of several repeated self-reports measure of perineal pain (each 4 hours) on an 11-point visual analogue scale (VAS) from 0 to 10.

SECONDARY OUTCOMES:
Rate of perineal laceration | 2 hours after delivery
  1st, 2nd, 3rd and 4th (OASIS) degree perineal lacerations
Rate of episiotomy | 2 hours after delivery
  episiotomy
Perineal healing assessed by the REEDA scale | 3 days after delivery
  Evaluation of perineal healing with the REEDA (redness, oedema, ecchymosis, discharge and approximation of the wound edges) scale: values from 0 to 15, higher scores meaning a worse perineal healing.
Change of perineal pain assessed by the VAS (<H96) | From delivery to 3 days after delivery
  Area under the curve of several repeated self-reports measure of perineal pain on an 11-point visual analogue scale (VAS) from 0 to 10.
Consumptions of pain relief medications | 3 days after delivery
  Number and type of pain relief medications consumed: paracetamol, nonsteroidal anti-inflammatory drugs, opioids, nefopam
Pain interference on daily functioning assessed by the BPI-SF | 2 months after delivery
  Pain interference on daily functioning assessed by the Brief pain inventory-short form scale (BPI-SF), 7 items from the subscale 23, each item independently scored from 0 to 10, higher score meaning higher pain interference on daily functioning.
Perineal complication | At two months postpartum
  Number of health care appointments (in or outpatient care) for perineal reason (general practitioner, midwife, obstetrician-gynaecologist …)
Childbirth experience assessed by the QACE | 3 days postpartum
  Childbirth experience assessed by the Short version of the Questionnaire for Assessing the Childbirth Experience (QACE). Scores for the 13 items range from 1-4 with higher scores indicating a more negative childbirth experience.
Rate of exclusive breastfeeding | At 3 days after delivery
  Breastfeeding as exclusive mode of infant feeding
Rate of exclusive breastfeeding | At 2 months after delivery
  Breastfeeding as exclusive mode of infant feeding
Rate of breastfeeding complications | At 2 months after delivery
  Breastfeeding complications reported by women : breast engorgement, mastitis, breast abscess
Urinary incontinence assessed with the ICIQ-UI SF | At 2 months after delivery
  Urinary incontinence assessed with the ICIQ - UI SF (International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form). Score ranges from 0 to 21, higher scores indicating higher urinary incontinence.
Anal incontinence assessed with the Wexner Score | At 2 months after delivery
  Anal incontinence assessed with the Wexner Score. Score ranges from 0 to 20, higher scores indicating higher anal incontinence.
Sexual function assessed with the FSFI | At 2 months after delivery
  Sexual function assessed by 4 items of the satisfaction et pain subscales of the FSFI (Female Sexual Function Index). Higher score for satisfaction (from 1 to 5) means higher satisfaction. Higher scores for pain items means higher pain (from 1 to 5).
Rate of postpartum depression assessed by the EPDS | At 2 months after delivery
  Postpartum depression assessed with the Edinburgh postnatal depression scale (EPDS). Score ranges from 0 to 30, higher scores meaning more depressive symptoms. Postpartum depression will be defined by a score greater than 12.

CONTACTS AND LOCATIONS:
Overall Officials: Anne CHANTRY, RM & PhD, Study Director — Assistance publique - Hôpitaux de Paris / INSERM
Locations (2):
- France (2):
  - Louis Mourier Hospital, Colombes
  - Cochin Hospital, Paris

IPD SHARING:
Plan to Share IPD: No